CLINICAL TRIAL: NCT00608387
Title: Web-based, Patient-centered Approach to CVD Risk-factor Management and Reduction
Brief Title: Evaluating a Web-Based Cardiovascular Disease Risk Factor Reduction Program Among American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills Center for American Indian Health (Other)
Collaborators: University of Washington (Other); University of Colorado, Denver (Other); NuMedics, Inc. (Industry); Cheyenne River Sioux Tribe Telephone Authority (Unknown); Missouri Breaks Industries Research, Inc. (Other); Cheyenne River Sioux Tribe (Other Government)
Responsible Party: Principal Investigator, Jeffrey Henderson, MD, MPH, President & CEO, Black Hills Center for American Indian Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 453; 1U01HL087422 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-02-06 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus, Type 2; Hypertension; Obesity; Tobacco Use Cessation
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Hypertension; Obesity; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Participants will receive usual care from their healthcare providers and have access to a Web-based CVD risk-factor management program.
  Interventions: Behavioral: Chronic disease management Web-based software
- B (No Intervention): Participants will receive usual care from their healthcare providers.

INTERVENTIONS:
Behavioral: Chronic disease management Web-based software — Participants will have access to remotely based medical providers through the use of the Web-based software.
  Other Names: CliniPro
  Arms: A

SUMMARY:
Cardiovascular disease (CVD) is a serious health concern for American Indians, but there have been few behaviorally based programs to lessen CVD risk among this population. The purpose of this study is to evaluate whether a Web-based program, in addition to usual medical care, can lower CVD risk factors among American Indians who have type 2 diabetes and a high risk of developing CVD.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of death among American Indians. Significant risk factors for CVD within the American Indian population include type 2 diabetes, tobacco use, poor dietary and physical activity habits, and poor medication and treatment adherence. Despite the fact that these risk factors can be reduced through behavior change, there have been few behaviorally based interventions aimed at American Indians to lessen their CVD risk. Research has shown that medical care is moving away from sporadic, standard doctors' office visits to a more continuous and interactive relationship with health care providers. A Web-based program that allows people to interact with remotely located doctors who can answer questions and provide advice may be beneficial at increasing treatment adherence and lowering CVD risk. This study will evaluate the use of a Web-based program at lowering CVD risk among American Indians with type 2 diabetes. Researchers will also analyze the cost-effectiveness of the Web-based program and the possible healthcare cost savings.

This 3-year study will enroll American Indian adults at high risk for CVD. Participants will be randomly assigned either to usual care at their local health facility or usual care plus the Web-based program. Participants using the Web-based program will have access to a Web site that will allow them to interact with two remotely based doctors. Participants will be able to send e-mail and instant messages to ask questions and receive information, advice, or motivational messages from the doctors. Participants will periodically enter their blood glucose test results and complete questionnaires online. Study visits, occurring twice a year for 3 years, will include blood pressure and body mass index (BMI) measurements, blood collection, and smoking status assessments.

ELIGIBILITY:
Inclusion Criteria:

* Completed a baseline Education and Research Towards Health (EARTH) study examination
* Diagnosed with type 2 diabetes mellitus AND hypertension and/or hyperlipidemia
* Able to read and understand English
* Able to walk

Exclusion Criteria:

* Diagnosed with CVD at study entry
* Currently receiving active treatment for any non-skin cell cancer
* Any medical condition that study physicians believe would interfere with study participation or evaluation of results
* Mental incapacity and/or cognitive impairment that would preclude adequate understanding of, or cooperation with, the study procedures
* Kidney insufficiency, as indicated by serum creatinine level greater than 2.0 mg/dL for women and greater than 2.4 mg/dL for men
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbgA1c) | Measured at Year 3

SECONDARY OUTCOMES:
Mean blood pressure | Measured at Year 3
Low-density lipoprotein cholesterol (LDL) | Measured at Year 3
BMI | Measured at Year 3
Smoking status | Measured at Year 3
Overall cost-effectiveness | Measured at Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Henderson, MD, MPH, Principal Investigator — Black Hills Center for American Indian Health
Locations (1):
- Black Hills Center for American Indian Health, Rapid City, South Dakota, United States

REFERENCES:
- [Background] Goldberg HI, Lessler DS, Mertens K, Eytan TA, Cheadle AD. Self-management support in a web-based medical record: a pilot randomized controlled trial. Jt Comm J Qual Saf. 2004 Nov;30(11):629-35, 589. doi: 10.1016/s1549-3741(04)30074-2. PMID 15565762
- [Background] Ralston JD, Revere D, Robins LS, Goldberg HI. Patients' experience with a diabetes support programme based on an interactive electronic medical record: qualitative study. BMJ. 2004 May 15;328(7449):1159. doi: 10.1136/bmj.328.7449.1159. PMID 15142919
- [Background] Goldberg HI, Ralston JD, Hirsch IB, Hoath JI, Ahmed KI. Using an Internet comanagement module to improve the quality of chronic disease care. Jt Comm J Qual Saf. 2003 Sep;29(9):443-51. doi: 10.1016/s1549-3741(03)29053-5. PMID 14513667
- [Background] Henderson JA, Chubak J, O'Connell J, Ramos MC, Jensen J, Jobe JB; LOWPK Project Team. Design of a randomized controlled trial of a web-based intervention to reduce cardiovascular disease risk factors among remote reservation-dwelling American Indian adults with type 2 diabetes. J Prim Prev. 2012 Aug;33(4):209-22. doi: 10.1007/s10935-012-0276-x. PMID 23001642